CLINICAL TRIAL: NCT02675959
Title: Safety and Efficacy of Prophylactic Defibrotide in Children, Adolescents, and Young Adults With Sickle Cell Disease or Beta Thalassemia Following MAC and Haploidentical Stem Cell Transplantation Utilizing CD34 Enrichment and T-Cell (CD3) Addback
Brief Title: Myeloablative Conditioning, Prophylactic Defibrotide and Haplo AlloSCT for Patients With Sickle Cell Disease
Acronym: NYMC-571
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Collaborators: University of California, Los Angeles (Other); Medical College of Wisconsin (Other); Tufts Medical Center (Other); Baylor College of Medicine (Other); Johns Hopkins University (Other); Dana-Farber Cancer Institute (Other); Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Mitchell Cairo, Principal Investigator, New York Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC 571; 4090 (Other Grant/Funding Number: OPD)
Record Dates: First submitted 2016-01-22; First posted 2016-02-05 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cell Disease
Keywords: stem cell transplantation; sickle cell disease; haploidentical; defibrotide
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — defibrotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Defibrotide prophylaxis (Experimental): defibrotide will be given prior to and during myeloablative immunotherapy conditioning (MAIC) followed by familial haploidentical (FHI) allogeneic stem cell transplantation (AlloSCT) with CD34 enrichment and t-cell addback in patients with high-risk sickle cell disease or beta thalassemia to reduced the risk and rate of the development of sinusoidal obstructive syndrome (SOS).
  Interventions: Drug: Defibrotide

INTERVENTIONS:
Drug: Defibrotide — defibrotide will be given prophylactically prior to AlloSCT to determine if it decreases the incidence of SOS in this high risk population, and determine that it is safe and feasible to give along with myeloimmunoablative therapy and allogeneic transplant.

SUMMARY:
This is a follow-up trial to NYMC 526 (NCT01461837) to assess the safety, efficacy and toxicity of administering Defibrotide prophylaxis for high-risk sickle cell or beta thalassemia patients undergoing a familial haploidentical allogeneic stem cell transplantation with CD34 enrichment and T-cell addback. This patient population historically has a risk of developing sinusoidal obstructive syndrome (SOS) and Defibrotide has demonstrated efficacy in treatment of SOS. The Funding Source is FDA OOPD.

ELIGIBILITY:
Inclusion Criteria:

* Disease: Homozygous Hemoglobin S Disease, or Hemoglobin S B0/+ thalassemia, or Hemoglobin SC Disease, or Beta thalassemia intermedia/majora
* Patients must demonstrate one or more of the following Sickle Cell Disease Complications (or patients in Cohort 2 can meet other high risk criteria instead)
* Clinically significant neurologic event (stroke) or any neurologic deficit lasting >24 hours that is accompanied by an infarct on cerebral MRI
* Acute chest syndrome in the preceding two year period prior to enrollment that have failed, been non-compliant or declined hydroxyurea treatment, or prior to chronic RBC transfusion therapy, exchange transfusion or erythrocyte pheresis.
* Recurrent painful events (at least 3 in the 2 years prior to enrollment or prior to chronic chronic RBC transfusion therapy, exchange transfusion or erythrocyte pheresis).
* Abnormal TCD study requiring starting on chronic transfusion therapy and/or exchange transfusions.
* At least one silent infarct lesion on a MRI scan of the head. Or (directly or probably related to SCD)
* Sickle Cell nephropathy;
* Splenic sequestration requiring RBC transfusion;
* Aplastic crisis requiring RBC transfusion;
* Avascular necrosis of the hip diagnosed by MRI;
* Two episodes or more of leg ulcerations;
* Recurrent priapism .
* Infant dactylitis.

  * OR for Cohort #2 ONLY: Patient must be between 18 and 34.99 years of age, patients must demonstrate at least two of the following:
* WBC > 13,500 cells/microliter at baseline when not acutely ill (on two separate occasions) > 2 weeks from a VOC event or hospitalization.
* Tricuspid Regurgitant Jet Velocity (TRV) > 3.0 m/s
* Requiring Chronic Monthly Transfusions ( > 12 transfusions in the 12 months)
* History of sepsis
* N-terminal pro-brain natriuretic peptide (NT-proBNP) > 160 ng/L at clinical baseline when not acutely ill or hospitalized.
* all patients must meet disease, age, organ function and donor criteria;

Exclusion Criteria:

* Patients who are receiving concomitant systemic anticoagulants and/or fibrinolytic therapies.
* Patients with a previously known hypersensitivity reaction to defibrotide.
* Females who are pregnant or breast-feeding are not eligible
* SCD Patients with documented uncontrolled infection at the time of study entry are not eligible.
* SCD patients who have an unaffected HLA matched family donor willing to proceed to donation will not be eligible for this study.
* Karnofsky or Lansky (age appropriate) Performance Score <50% (hemiplegia alone secondary to a previous stroke is not an exclusion)
* Demonstrated lack of compliance with medical care.
* Patients with clinically significant fibrosis or cirrhosis of the liver will not be eligible.
* Patients who have previously received a HSCT will not be eligible.
* Patients with contraindications to the use of defibrotide

Ages: 6 Months to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
All patients will be monitored for known and unknown side effects of defibrotide with daily physical exams while in the hospital and then as needed in addition to daily laboratory values including chemistries, hematology labs as needed | 100 days
  Patients will be given Defibrotide prophylaxis starting 10 days before the stem cell infusion at 6.25 mg/kg IV q6h and continue through Day +21.
All patients will be monitored for the development of SOS. | 1 year
  All patients will get daily lab values while in patients and then as needed to monitor for elevation in liver function tests and other abnormal chemistry or hematology values. Imaging on the liver will be performed as needed to determine if they develop SOS with defibrotide.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cairo, MD, Principal Investigator — New York Medical College
Locations (4):
- United States (4):
  - University of California Los Angeles, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - New York Medical College, Valhalla, New York
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chu Y, Talano JA, Baxter-Lowe LA, Verbsky JW, Morris E, Mahanti H, Ayello J, Keever-Taylor C, Johnson B, Weinberg RS, Shi Q, Moore TB, Fabricatore S, Grossman B, van de Ven C, Shenoy S, Cairo MS. Donor chimerism and immune reconstitution following haploidentical transplantation in sickle cell disease. Front Immunol. 2022 Dec 9;13:1055497. doi: 10.3389/fimmu.2022.1055497. eCollection 2022. PMID 36569951